CLINICAL TRIAL: NCT03536962
Title: Cohort Study: Multidisciplinary Follow-up of Patients With Amyotrophic Lateral Sclerosis
Brief Title: Multidisciplinary Follow-up of Patients With Amyotrophic Lateral Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ruxandra Iancu Ferfoglia (Other)
Responsible Party: Sponsor-Investigator, Ruxandra Iancu Ferfoglia, Chief resident, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: NAC 11-062R
Record Dates: First submitted 2018-01-14; First posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Analyse a multidisciplinary follow-up of amyotrophic lateral sclerosis patients, monitored through a Cohort study at Geneva University Hospitals.

DETAILED DESCRIPTION:
Since April 2010 a quarterly follow-up is available for patients with ALS at Geneva University Hospitals. It takes place in the outpatient unit of the Department of Neurology, and includes interventions by the multidisciplinary team of the " Center for Amyotrophic Lateral Sclerosis and related diseases ". This new tracking method can help improving quality of life of patients and their families by adapting medical care, proposing communication aids, facilitating access to specialized examinations and anticipating pulmonary, nutritional and neurologic complications. Moreover, it speeds up administrative procedures, improves the flow of information between medical teams inside and outside the hospital and it allows and encourages discussion about advanced directives.

Since June 2012, the multidisciplinary follow-up is monitored through a Cohort study that was approved by the ethical committee (NAC 11-062R). We collect clinical examination findings, anthropometric evaluation, blood analyses, pulmonary function tests, respiratory muscle strength, arterial blood gases, nocturnal oximetry, and evaluation by occupational therapists and by physiotherapists on a quarterly basis. Nerve conduction studies are done at the beginning of the follow-up to identify the degree and extent of loss of upper and lower motoneurons in ALS and to help guiding the diagnosis. MRI and analysis of cerebrospinal fluid are also acquired at the beginning of the follow-up in order to rule out other diagnoses which can mimic ALS. Definite, probable or possible ALS is defined according to the Revised El Escorial and Awaji criteria [16-17]. Patients are referred to a genetic counselor who helps making informed decisions regarding genetic issues. The data collected are inserted into the Secu-Trial database, which is managed by an assistant provided by the Clinical Research Center.

ELIGIBILITY:
Inclusion Criteria:

Amyotrophic Lateral Sclerosis fulfilling the El Escorial criteria (definite, probable, possible), primary lateral sclerosis, progressive muscular atrophy, progressive bulbar palsy

Exclusion Criteria:

Patients with other neurological diagnoses than mentioned in the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients living in the Geneva area suffering from Amyotrophic Lateral Sclerosis or related disorders
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal change of the revised Amyotrophic Lateral Sclerosis Functional rating scale in Amyotrophic Lateral Sclerosis patients | 2012-2016
  Clinical evolution of Amyotrophic Lateral Sclerosis patients will be measured by the revised Amyotrophic Lateral Sclerosis Functional rating scale. This scale includes 12 questions covering 4 distinct domains: fine motor function, gross motor function, respiratory function and bulbar symptoms. Lower scores indicate higher disability.This score will be assessed every three months

SECONDARY OUTCOMES:
Correlation of walking speed measured by Timed Up and Go test and the Amyotrophic Lateral Sclerosis Functional rating scale (ALSFRS-R) | 2012-2016
  the Timed Up and Go test measures the time needed to rise from a chair walk 3 m, turn around and return to a seated position. The speed at which patients perform this test is measured in seconds and will be assessed at each trimestrial visit and will be correlated the (ALSFRS-R)
Longitudinal evolution of pulmonary function in ALS patients | 2012-2016
  Vital capacity(in Liters) will be assessed at each trimestrial visit
Evolution of body mass composition measured by the Body Mass Index in ALS patients | 2012-2016
  the Body Mass Index (kg/m2), will be assessed at each trimestrial visit
Longitudinal evolution of inspiratory muscle strength in ALS patients | 2012-2016
  inspiratory muscle strength (in cmH2O) will be assessed at each trimestrial visit

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Janssens, MD, Study Chair — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to multidisciplinary consultation for motorneurone disease — http://www.hug-ge.ch/neurologie/centre-sla